CLINICAL TRIAL: NCT06978153
Title: Perioperative Treatment With Benmelstobart Combined With Chemotherapy With or Without Anlotinib in Resectable Limited-Stage Small Cell Lung Cancer: A Randomized, Two-Cohort, Multicenter, Phase II Clinical Study
Brief Title: This is a Two-cohort, Exploratory Clinical Study Assessing the Activity of Benmelstobart Combined With Chemotherapy With or Without Anlotinib in Resectable Limited-Stage Small Cell Lung Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Shaanxi-Lung-03
Record Dates: First submitted 2025-05-10; First posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Limited Stage Small Cell Lung Cancer
MeSH Terms: interventions — Drug Therapy; anlotinib

STUDY DESIGN:
Intervention Model Description: Model Description
Masking Description: Masking Description
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1: Neoadjuvant therapy (benmelstobart combined with chemotherapy and anlotinib) (Experimental): Cohort 1: Neoadjuvant therapy (benmelstobart combined with chemotherapy and anlotinib, 3 cycles, every 21 days is a cycle) : benmelstobart, 1200mg, iv, day 1. Anlotinib, 10 mg, po, qd, was taken orally for 2 consecutive weeks and stopped for 1 week. Anlotinib was stopped 1 week before surgery. Etoposide, 100mg/m2, day 1~3. Cisplatin, 75mg/m2，day 1; or Carboplatin, AUC 5, day 1. Surgery was performed 4-6 weeks after the final administration of benmelstobart as assessed by the investigator. Adjuvant therapy was evaluated by the investigator 4-6 weeks after surgery. Patients who achieved R0 resection received adjuvant therapy (benmelstobart combined with anlotinib, 12 cycles, every 21 days is a cycle) : benmelstobart, 1200mg, iv, day1; anlotinib, 10 mg, po, qd, was taken orally for 2 weeks and stopped for 1 week.
  Interventions: Drug: benmelstobart combined with chemotherapy and anlotinib
- Cohort 2: Neoadjuvant therapy (benmelstobart combined with chemotherapy) (Experimental): Cohort 2: Neoadjuvant therapy (benmelstobart combined with chemotherapy, 3 cycles, every 21 days is a cycle) : benmelstobart, 1200mg, iv, day1; Etoposide, 100mg/m2, day 1~3; Cisplatin, 75mg/m2，day 1; or Carboplatin, AUC 5, day 1. Surgery was performed 4-6 weeks after the final administration of benmelstobart as assessed by the investigator. Adjuvant therapy was evaluated by the investigator 4-6 weeks after surgery. Patients who achieved R0 resection received adjuvant therapy (benmelstobart, every 21 days is a cycle) : benmelstobart, 1200mg, iv, day1.
  Interventions: Drug: benmelstobart combined with chemotherapy

INTERVENTIONS:
Drug: benmelstobart combined with chemotherapy and anlotinib — Cohort 1: Neoadjuvant therapy (benmelstobart combined with chemotherapy and anlotinib, 3 cycles, every 21 days is a cycle) : benmelstobart, 1200mg, iv, day 1. Anlotinib, 10 mg, po, qd, was taken orally for 2 consecutive weeks and stopped for 1 week. Anlotinib was stopped 1 week before surgery. Etoposide, 100mg/m2, day 1~3. Cisplatin, 75mg/m2，day 1; or Carboplatin, AUC 5, day 1. Surgery was performed 4-6 weeks after the final administration of benmelstobart as assessed by the investigator. Adjuvant therapy was evaluated by the investigator 4-6 weeks after surgery. Patients who achieved R0 resection received adjuvant therapy (benmelstobart combined with anlotinib, 12 cycles, every 21 days is a cycle) : benmelstobart, 1200mg, iv, day1; anlotinib, 10 mg, po, qd, was taken orally for 2 weeks and stopped for 1 week.
  Arms: Cohort 1: Neoadjuvant therapy (benmelstobart combined with chemotherapy and anlotinib)
Drug: benmelstobart combined with chemotherapy — Cohort 2: Neoadjuvant therapy (benmelstobart combined with chemotherapy, 3 cycles, every 21 days is a cycle) : benmelstobart, 1200mg, iv, day1; Etoposide, 100mg/m2, day 1~3; Cisplatin, 75mg/m2，day 1; or Carboplatin, AUC 5, day 1. Surgery was performed 4-6 weeks after the final administration of benmelstobart as assessed by the investigator. Adjuvant therapy was evaluated by the investigator 4-6 weeks after surgery. Patients who achieved R0 resection received adjuvant therapy (benmelstobart, every 21 days is a cycle) : benmelstobart, 1200mg, iv, day1.
  Arms: Cohort 2: Neoadjuvant therapy (benmelstobart combined with chemotherapy)

SUMMARY:
A total of 66 patients were enrolled in this exploratory study and randomly assigned to cohort 1 and cohort 2, with 33 patients in each group. Cohort 1: Neoadjuvant therapy (benmelstobart combined with chemotherapy and anlotinib, 3 cycles, every 21 days is a cycle). Surgery was performed 4-6 weeks after the final administration of benmelstobart as assessed by the investigator. Adjuvant therapy was evaluated by the investigator 4-6 weeks after surgery. Patients who achieved R0 resection received adjuvant therapy (benmelstobart combined with anlotinib, 12 cycles, every 21 days is a cycle). Cohort 2: Neoadjuvant therapy (benmelstobart combined with chemotherapy, 3 cycles, every 21 days is a cycle). Surgery was performed 4-6 weeks after the final administration of benmelstobart as assessed by the investigator. Adjuvant therapy was evaluated by the investigator 4-6 weeks after surgery. Patients who achieved R0 resection received adjuvant therapy (benmelstobart, every 21 days is a cycle) .

ELIGIBILITY:
Inclusion Criteria:

* Patients voluntarily participate in this study, sign the informed consent form, demonstrate good compliance, and cooperate with follow-up.
* Aged 18 to 75 years (inclusive) at the time of signing informed consent, regardless of gender.
* Histologically confirmed small cell lung cancer (SCLC).
* Confirmed as stage I-IIIB SCLC (T1-3N0-2M0) per AJCC 9th Edition.
* Patients who have received 1 cycle of chemotherapy are eligible; no other prior treatments are permitted.
* ECOG Performance Status (PS) 0 or 1.
* Assessed by the investigator as having no surgical contraindications.
* At least one measurable lesion per RECIST 1.1 criteria.
* Expected survival ≥8 weeks.
* Women of childbearing potential (aged 15-49) must have a negative serum pregnancy test within 7 days before treatment initiation and agree to use reliable contraception during the study until 8 weeks after discontinuation. Normal function of major organs meeting the following criteria:
* Hematologic tests (no blood transfusion, blood products, G-CSF, or hematopoietic stimulants within 14 days): Hemoglobin (Hb) ≥90 g/L; Absolute neutrophil count (ANC) ≥1.5×10⁹/L; Platelets (PLT) ≥80×10⁹/L.
* Biochemical tests meeting: Total bilirubin (TBIL) ≤1.5×ULN; ALT/AST ≤2.5×ULN; Serum creatinine (Cr) ≤1.5×ULN or creatinine clearance (CCr) ≥60 mL/min.
* Urine protein <2+; for patients not on anticoagulation: INR ≤1.5, APTT ≤1.5×ULN. Patients on full-dose or parenteral anticoagulants may enroll if dosing has been stable for ≥2 weeks and coagulation tests are within therapeutic ranges.

Exclusion Criteria:

* Histologically confirmed mixed-type SCLC.
* Extensive-stage SCLC.
* ECOG PS >1.
* Active or untreated CNS metastases confirmed by CT/MRI during screening/prior imaging.
* Uncontrolled tumor-related pain.
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage (≥1×/month).
* Uncontrolled/symptomatic hypercalcemia (ionized calcium >1.5 mmol/L, calcium >12 mg/dL, or corrected serum calcium >ULN).
* Systemic immunostimulants (e.g., IFN-α, IL-2, TNF) within 4 weeks prior to enrollment (cancer vaccines allowed if prior).
* Systemic corticosteroids (>10 mg prednisone/day or equivalent) or immunosuppressants within 14 days, except: Replacement therapy (≤10 mg prednisone/day); Topical/ocular/intra-articular/nasal/inhaled steroids with minimal systemic absorption; Short-term (≤7 days) prophylactic use (e.g., contrast allergy) or for non-autoimmune conditions.
* Imaging-confirmed tumor invasion of major vessels or high risk of fatal hemorrhage per investigator; or cavitary/necrotic lung tumors.
* Other malignancies within 5 years except: cervical CIS, cured basal cell carcinoma, Ta/Tis bladder tumors.
* Prior use of anlotinib or other antiangiogenic agents.
* Prior anti-PD-1/PD-L1/CTLA-4 antibodies or other T-cell co-stimulation/checkpoint pathway therapies (e.g., ICOS, CD40/CD137/GITR/OX40 agonists).
* Hypersensitivity to anlotinib or benmelstobart components.
* Factors impairing oral drug intake (e.g., dysphagia, chronic diarrhea, intestinal obstruction).
* Uncontrolled comorbidities including:

  1. Poorly controlled hypertension (SBP ≥150 mmHg, DBP ≥100 mmHg);
  2. Grade ≥1 myocardial ischemia/infarction, arrhythmias (QTc ≥480 ms), or ≥NYHA Class II heart failure;
  3. Abnormal coagulation (INR >1.5, PT >ULN+4s, APTT >1.5×ULN), bleeding tendency, or thrombolytic/anticoagulant therapy (prophylactic low-dose heparin [6,000-12,000 U/day] or aspirin [≤100 mg/day] allowed if INR ≤1.5);
  4. Active/severe uncontrolled infections;
  5. Cirrhosis, decompensated liver disease, active/chronic hepatitis requiring antivirals;
  6. Renal failure requiring dialysis;
  7. Immunodeficiency (HIV+, congenital/acquired immunodeficiency) or organ transplant history;
  8. Poorly controlled diabetes (FBG >10 mmol/L);
  9. Urine protein ≥++ or 24-h urine protein >1.0 g;
  10. Epilepsy requiring treatment;
  11. Non-healing wounds/fractures.
* Significant hemoptysis (>50 mL/day within 2 weeks) or clinically significant bleeding (e.g., GI bleeding, hemorrhagic gastric ulcer, baseline fecal occult blood ≥++).
* Interstitial lung disease (ILD), drug-induced ILD, steroid-requiring radiation pneumonitis, or active ILD.
* Arterial/venous thromboembolism within 6 months (e.g., stroke [including TIA], DVT, PE).
* Grade ≥2 peripheral neuropathy (excluding trauma-related).
* Major surgery/severe trauma with residual effects within 14 days.
* Concurrent clinical trials or <4 weeks from prior trial treatment.
* Live/attenuated vaccination within 30 days before benmelstobart or planned during study.
* History of severe hypersensitivity to monoclonal antibodies.
* Pregnant/lactating women.
* Uncontrolled psychiatric/neurological disorders affecting compliance.
* Other factors per investigator judgment that may lead to study termination (e.g., severe illness, lab abnormalities, or social/family constraints compromising safety/data collection).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-05-20 (Estimated); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
event-free survival (EFS) | up to 2 years
  The event-free survival (EFS) is defined as the duration from randomization to the occurrence of any event, which includes disease progression, postoperative recurrence, discontinuation of treatment for any reason, or death.

SECONDARY OUTCOMES:
Major pathologic response rate (MPR) | 7 days after surgery
  Major pathologic response rate (MPR) as assessed/estimated by the investigator, i.e. the proportion of residual surviving tumor cells in the tumor bed in the postoperative specimen ≤10%
Complete pathological response (pCR) | 7 days after surgery
  Complete pathological response (pCR): defined as no residual tumor cells in postoperative tumor tissue specimens (including no tumor residue in lymph nodes), based on pathological response
Objective response rate (ORR) | 7 days after surgery
  The proportion of patients who exhibit a partial response (PR) or complete response (CR) to treatment is defined as follows.
overall survival (OS) | up to 3 year
  Overall survival (OS) refers to the duration from the initiation of randomization until death occurs for any reason.
Treatment-related adverse events evaluated according to CTCAE v5.0 | up to 2 years
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0
Surgical complications evaluated according to the Clavien-Dindo classification | up to 2 years
  Number of participants with surgical complications as assessed by Clavien-Dindo

IPD SHARING:
Plan to Share IPD: No